CLINICAL TRIAL: NCT06695091
Title: Clinical Assessment of Endodontically Treated Posterior Teeth Prepared With Two Occlusal Designs and Two Ceramic Full Coverage Restorations (Randomized Clinical Trial)
Brief Title: Clinical Assessment of Endodontically Treated Posterior Teeth Prepared With Two Occlusal Designs and Two Ceramic Full Coverage Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Abou-steit, Lecturer of fixed prosthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-2020-9-120
Record Dates: First submitted 2022-11-29; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Clinical Behavioral
Keywords: Lithium disilicate; Zirconia; All-ceramic crowns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Triple blinded: The trial participants, the outcome assessors and the data analysis statistician are blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flat occlusal scheme (Active Comparator): occlusal design
  Interventions: Procedure: Monolithic zirconia crown; Procedure: Monolithic lithium disilicate crown
- Anatomic occlusal scheme (Active Comparator): occlusal design
  Interventions: Procedure: Monolithic zirconia crown; Procedure: Monolithic lithium disilicate crown

INTERVENTIONS:
Procedure: Monolithic zirconia crown — All-ceramic crown
Procedure: Monolithic lithium disilicate crown — All-ceramic crown

SUMMARY:
The aim of this study was to assess the impact of flat occlusal preparation design (FOD) of endodontically treated molars on the fracture resistance and distribution of stresses among a ceramic crown-molar structure when compared to two planes occlusal preparation design (TOD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with posterior root canal treated teeth that require full coverage restoration.
* 20 - 50 years old.
* Males or Females.
* Good oral hygiene.
* Presence of favorable occlusion and teeth are in normal alignment with the adjacent teeth.
* Patients agreed to return to follow-up evaluation.

Exclusion Criteria:

* Active periodontal or pulpal diseases.
* Lack of opposing dentition.
* Severe medical complications.
* Pregnancy.
* Lack of compliance.
* Evidence of parafunctional habits
* Temporomandibular joint disorders

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Fracture | 12 months
  Using Modified United States Public Health Service (USPHS) criteria

SECONDARY OUTCOMES:
Marginal adaptation | 12 months
  Using Modified United States Public Health Service (USPHS) criteria
Marginal discoloration | 12 months
  Using Modified United States Public Health Service (USPHS) criteria
Secondary caries | 12 months
  Using Modified United States Public Health Service (USPHS) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Abou-Steit, Lecturer, Principal Investigator — Lecturer of Fixed Prosthodontics
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Mannocci F, Cowie J. Restoration of endodontically treated teeth. Br Dent J. 2014 Mar;216(6):341-6. doi: 10.1038/sj.bdj.2014.198. PMID 24651340
- [Background] Varlan C, Dimitriu B, Varlan V, Bodnar D, Suciu I. Current opinions concerning the restoration of endodontically treated teeth: basic principles. J Med Life. 2009 Apr-Jun;2(2):165-72. PMID 20108535
- [Background] Beier US, Kapferer I, Dumfahrt H. Clinical long-term evaluation and failure characteristics of 1,335 all-ceramic restorations. Int J Prosthodont. 2012 Jan-Feb;25(1):70-8. PMID 22259801
- [Background] Nagasiri R, Chitmongkolsuk S. Long-term survival of endodontically treated molars without crown coverage: a retrospective cohort study. J Prosthet Dent. 2005 Feb;93(2):164-70. doi: 10.1016/j.prosdent.2004.11.001. PMID 15674228
- [Background] Oyar P, Ulusoy M, Eskitascioglu G. Finite element analysis of stress distribution in ceramic crowns fabricated with different tooth preparation designs. J Prosthet Dent. 2014 Oct;112(4):871-7. doi: 10.1016/j.prosdent.2013.12.019. Epub 2014 Apr 21. PMID 24750896